CLINICAL TRIAL: NCT05886127
Title: Treatment of Immediate and Prevention of Delayed Bleeding After Endoscopic Retrograde Cholangiopancreatography Sphincterothomy or Precut With a Novel Self-assembling Peptide Hemostatic Gel. A Single Centre Prospective Observational Nonrandomized Study
Brief Title: Treatment of Postsphincterotomy Bleeding With a Novel Self-assembling Peptide Hemostatic Gel.
Acronym: ERCPURA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Petr Hrabak, Principal investigator, General University Hospital, Prague
Other Study IDs: ERCP-PURA/1
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Biliary Obstruction; Complication of Treatment
Keywords: ERCP; A novel haemostatic agent; Postsfincterothomy bleeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients undergoing ERCP with papilosphincterotomy or precut: All patients after ERCP papilosphincterotomy or precut will receive a novel hemostatic agent (Purastat®)
  Interventions: Device: A novel hemostatic agent (Purastat®)
- Historical control: All patients who had ERCP with papilosphincterotomy or precut in the previous period, when a novel hemostatic gel (Purastat®) was not available.

INTERVENTIONS:
Device: A novel hemostatic agent (Purastat®) — A novel hemostatic agent (Purasta®) will be applied on cutted ampulla of Vater
  Groups: Patients undergoing ERCP with papilosphincterotomy or precut

SUMMARY:
The aim of this observational study is to evaluate safety and efficacy of a novel self-assembling peptide hemostatic gel in reduction of bleeding after endoscopic sphincterotomy during ERCP (endoscopic retrograde cholangiopancreatography )

DETAILED DESCRIPTION:
ERCP with sfincterotomy or precut is connected with procedural or/and postprocedural bleeding. Estimated risk of bleeding is from 2% to 10%. Procedural bleeding is usually managed by diluted epinephrine injection, balloon tamponade, hemoclip or fully covered metalic self-expanding stent placement. There is no standard preventive treatment for patients with higher risk of delayed post-sphincterotomy bleeding. PuraStat®, 3D Matrix Europe SAS, Caluire-et-Cuire, France) is synthetic self-assembling peptide haemostatic gel indicated to stop bleeding from small blood vessel or oozing from capillaries. Purastat® is easily aplicated through a catheter during the ERCP procedure and it is not significantly prolonging the procedure. The transparent gel is not compromising the endoscopic view and enables to continue in procedure if necessary.

All patients after ERCP sfincterotomy or precut will recieve Purastat® during the procedure Adverse events (bleeding, cholangoitis, pancreatitis) will be monitored during following 4 weeks (ambulatory after hospital discharge) This cohort will be compared to historical control, when Purastat® was not available tu use.

ELIGIBILITY:
Inclusion Criteria:

* . All patients indicated for ERCP with papilosphincterotomy or precut.
* Participant is willing and able to give informed consent for participation in the study

Exclusion Criteria:

* Known allergy to a novel hemostatic agent
* Gravidity
* Inability to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients indicated for ERCP with sphincterotomy or precut at our endoscopy centre. Patients are mostly reffered from adjacent territory belonging to our hospital (non-selected cohort)
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of bleeding episodes after ERCP sfincterothomy or precut | One month

SECONDARY OUTCOMES:
Number of nonbleeding complications after ERCP sfincterothomy or precut | One month

CONTACTS AND LOCATIONS:
Overall Officials: Petr Hrabak, Principal Investigator — General University Hospital, Prague
Locations (1):
- Petr Hrabak, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
The results will be presented at Czech and Slovak gastroenterology meeting conference 2023 and in a peer-review journal.
Supporting Information: CSR
Time Frame: We expect the availibility of CSR at the beginning of 2024 and will be available for 3 years
Access Criteria: The results will be available on request.

REFERENCES:
- [Background] Cotton PB, Lehman G, Vennes J, Geenen JE, Russell RC, Meyers WC, Liguory C, Nickl N. Endoscopic sphincterotomy complications and their management: an attempt at consensus. Gastrointest Endosc. 1991 May-Jun;37(3):383-93. doi: 10.1016/s0016-5107(91)70740-2. PMID 2070995
- [Background] Subramaniam S, Kandiah K, Chedgy F, Fogg C, Thayalasekaran S, Alkandari A, Baker-Moffatt M, Dash J, Lyons-Amos M, Longcroft-Wheaton G, Brown J, Bhandari P. A novel self-assembling peptide for hemostasis during endoscopic submucosal dissection: a randomized controlled trial. Endoscopy. 2021 Jan;53(1):27-35. doi: 10.1055/a-1198-0558. Epub 2020 Jul 17. PMID 32679602
- [Background] de Nucci G, Reati R, Arena I, Bezzio C, Devani M, Corte CD, Morganti D, Mandelli ED, Omazzi B, Redaelli D, Saibeni S, Dinelli M, Manes G. Efficacy of a novel self-assembling peptide hemostatic gel as rescue therapy for refractory acute gastrointestinal bleeding. Endoscopy. 2020 Sep;52(9):773-779. doi: 10.1055/a-1145-3412. Epub 2020 Apr 21. PMID 32316041
- [Background] Lin WC, Lin HH, Hung CY, Shih SC, Chu CH. Clinical endoscopic management and outcome of post-endoscopic sphincterotomy bleeding. PLoS One. 2017 May 17;12(5):e0177449. doi: 10.1371/journal.pone.0177449. eCollection 2017. PMID 28545082
- [Background] Tsou YK, Lin CH, Liu NJ, Tang JH, Sung KF, Cheng CL, Lee CS. Treating delayed endoscopic sphincterotomy-induced bleeding: epinephrine injection with or without thermotherapy. World J Gastroenterol. 2009 Oct 14;15(38):4823-8. doi: 10.3748/wjg.15.4823. PMID 19824118